CLINICAL TRIAL: NCT01545570
Title: A Single-blinded, Randomized, Placebo-controlled, Staggered-parallel, Escalating Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK2374697 in Healthy Volunteers
Brief Title: A Study to Determine the Safety, Tolerability, and Effects of GSK2374697 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114403
Record Dates: First submitted 2011-11-03; First posted 2012-03-06 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2376497 (Active Comparator): single dose escalation or multiple-dose titration
  Interventions: Drug: GSK2376497
- 0.9% sodium chloride (Placebo Comparator): placebo injection
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: GSK2376497 — GSK2376497 Active Comparator
  Arms: GSK2376497
Drug: 0.9% sodium chloride — 0.9% sodium chloride Placebo Comparator
  Arms: 0.9% sodium chloride

SUMMARY:
This is a single-blinded, randomized, placebo-controlled, staggered-parallel, escalating dose study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of GSK2374697 in healthy volunteers. The study will enrol approximately 72 subjects at one clinical study center in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and Holter monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included if the investigator and the GSK Medical Monitor (or designee) agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or objectives. Subjects with values outside the ranges noted below should be excluded from enrollment, unless the investigator and GSK medical monitor (or designee) agree that the value in question would not pose a significant safety risk for the subject or compromise the study objectives. Please see Section 7.1 for additional information.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2- 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study.

* Body weight ≥ 50.0 kg and BMI within the range 19.9 - 35 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Single or Average QTcB < 450 msec.
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN at screening and at baseline (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of chronic or acute pancreatitis. Note: Subjects with a lipase value above the upper limit of normal (ULN) at screening are excluded. If amylase result is above ULN and lipase is below ULN, an amylase isoenzyme analysis may be performed. If this additional test confirms that the pancreatic amylase isoenzyme fraction is not the cause of the elevation, the subject may enroll in the study.
* History of thyroid disease: personal or family history of thyroid cancer unless approved by the GSK medical monitor (or designee), and/or a history of uncorrected thyroid dysfunction or an abnormal thyroid function as assessed by TSH, and/or plasma calcitonin at screening > 50pg/mL.
* History of- or family history of a renal disorder that may compromise renal function
* Creatinine clearance < 80 mL/min. (estimated from serum creatinine (SCr) and demographic data using the Cockcroft-Gault calculation):

To calculate estimated Cockcroft-Gault GFR (mL/min) manually:

= (140 - age) * (weight in kg) * (0.85 if female) / (72 * Cr in mg/dL)

* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.

* Exposure to more than four new chemical entities within 12 months prior to the first dosing day, and prior exposure to any anti-diabetic drug in a clinical study will require approval from the GSK medical monitor (or designee) before a subject is considered eligible for enrollment. In addition, subject has participated in a clinical trial and has received an investigational (non-approved) product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor (or designee), contraindicates their participation. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and GSK Medical Monitor (or designee) the medication will not interfere with the study procedures or compromise subject safety.
* Where participation in the study would result in donation of blood or blood products in excess of approximately 500 mL within a 56 day period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-11-07 (Actual); Primary Completion 2012-12-23 (Actual); Study Completion 2012-12-23 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events after ascending single or titrated mulitple subcutaneous doses of GSK2374697 | up to 70 days post dose
  Adverse events, laboratory parameters, ECGs, and vital signs
pharmacokinetic parameters of GSK2374697, after ascending single or titrated multiple subcutaneous doses, in healthy subjects | pre-dose, then 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, and 66 hours after dose (this schedule is q6h through Day 3, up to just prior to Day 4). In addition, sampling continues out through Day 70, on specific days, q12h.
  Pharmacokinetics parameters: AUCs, Cmax, tmax, elimination half-life (t½), lag time (tlag), apparent clearance (CL/F) and apparent volume of distribution (V/F), area under the plasma drug concentration versus time curve on Days 1 through end of study (up to 70 Days)

SECONDARY OUTCOMES:
pharmacodynamic effects of GSK2374697 in healthy subjects after meal challenge | On 2 days
  Fasting, 2h, and Cmax parameters on Day -1 and approximately Day 6 (or Day 16)
dose proportionality of GSK2374697 | up to 70 days post dose
  Pharmacokinetics parameters based on single and/or titrated multiple subcutaneous doses of GSK2374697

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lin J, Hodge RJ, O'Connor-Semmes RL, Nunez DJ. GSK2374697, a long duration glucagon-like peptide-1 (GLP-1) receptor agonist, reduces postprandial circulating endogenous total GLP-1 and peptide YY in healthy subjects. Diabetes Obes Metab. 2015 Oct;17(10):1007-10. doi: 10.1111/dom.12533. Epub 2015 Aug 11. PMID 26179090
- See also: Results for study 114403 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114403?search=study&search_terms=114403#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register